CLINICAL TRIAL: NCT05182554
Title: Increasing the Effectiveness and Diffusion of COVID-19 Messaging for Vaccination
Brief Title: COVID-19 Messaging for Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Collaborators: Facebook, Inc. (Other); Code3 (Industry); Stanford University (Other); Harvard University (Other); Yale University (Other); Johns Hopkins University (Other); Massachusetts General Hospital (Other); Ludwig-Maximilians - University of Munich (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2106000397
Record Dates: First submitted 2021-10-21; First posted 2022-01-10 (Actual); Results first posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Vaccination Refusal; COVID-19 Pandemic
Keywords: Covid-19 Vaccine; Social Media
MeSH Terms: conditions — Vaccination Refusal; COVID-19

STUDY DESIGN:
Intervention Model Description: There are four arms in the study which geographic areas are assigned to in parallel. The geographic areas in the three treatment arms will receive a Facebook ad campaign over the same time period to one another.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): No intervention in this arm; the study team will examine publicly available county- and zip code-level outcomes in this group.
- Treatment 1: Direct (Experimental): Facebook users in the area receive ads which include videos of health professionals telling them to get vaccinated. The health professionals answer common questions about Covid-19 vaccines (e.g. are they safe / are they free).
  Interventions: Behavioral: Doctor Videos
- Treatment 2: Friends (Experimental): Facebook users in the area receive ads which include videos of health professionals encouraging them to help their friends to get vaccinated. There is also a link in the ad to a website build by the study team. This website hosts videos which answer common questions about vaccination (the same videos which are directly served to Facebook users in Treatment 1).
  Interventions: Behavioral: Doctor Videos; Behavioral: Sharing Videos; Behavioral: Vaccine Ambassador; Behavioral: Video framing; Behavioral: Video order
- Treatment 3: Gossips (Experimental): Facebook users in the area receive ads which include videos of health professionals encouraging them to nominate their most influential friends to help their friends get vaccinated. The difference from Treatment 2 is that the health professionals call on Facebook users to get their most influential friends to do the convincing about the vaccine. There is also a link in the ad to a website built by the study team. This website hosts videos which answer common questions about vaccination (the same videos that are directly served to Facebook users in Treatment 1).
  Interventions: Behavioral: Doctor Videos; Behavioral: Sharing Videos (Influencers); Behavioral: Vaccine Ambassador; Behavioral: Video framing; Behavioral: Video order

INTERVENTIONS:
Behavioral: Doctor Videos — Receive ads on Facebook or through our website with videos in which health professionals tell people to get the Covid-19 vaccine. The health professionals answer common questions about the Covid-19 vaccine, such as how mRNA vaccines work, and what types of side effects to expect.
  Arms: Treatment 1: Direct; Treatment 2: Friends; Treatment 3: Gossips
Behavioral: Sharing Videos — Receive ads on Facebook with videos in which health professionals tell people to encourage their unvaccinated friends to get the Covid-19 vaccine.
  Arms: Treatment 2: Friends
Behavioral: Sharing Videos (Influencers) — Receive ads on Facebook with videos in which health professionals tell people to get their most influential friends to encourage their unvaccinated friends to get the Covid-19 vaccine.
  Arms: Treatment 3: Gossips
Behavioral: Vaccine Ambassador — Adults in participating geographic areas can sign up to be a "vaccine ambassador" on a website that the study team has built. The study team will send updates to vaccine ambassadors when new content has been posted to the website (e.g. a new video) and/or to remind the vaccine ambassadors to encourage their friends to get vaccinated. The study team will incentivize vaccine ambassadors by entering participating ambassadors into a lottery for a prize.
  Arms: Treatment 2: Friends; Treatment 3: Gossips
Behavioral: Video framing — The same videos will be displayed using two different frames: a "myth" frame and a "fact" frame. Visitors to the vaccine content website will randomly receive one framing of each video.
  Arms: Treatment 2: Friends; Treatment 3: Gossips
Behavioral: Video order — The order in which videos appear on the vaccine content website will be randomized.
  Arms: Treatment 2: Friends; Treatment 3: Gossips

SUMMARY:
This study will distribute videos of health professionals encouraging Covid-19 vaccination to a large sample of Facebook users, and will test the most effective ways to maximize diffusion of this vaccine-related content to increase vaccination rates. The study sample will be U.S. states where vaccination rates remained low in fall 2021. The experimental design is an RCT with 4 groups, randomized at the county level: 1) a control group which receives no intervention, 2) a treatment group in which Facebook users receive ads which include videos of health professionals telling them to get vaccinated, 3) a treatment group in which Facebook users receive ads which include videos of health professionals encouraging them to help their friends to get vaccinated, and 4) a treatment group in which Facebook users receive ads which include videos of health professionals encouraging them to get their most influential friends to help their friends get vaccinated. In treatments 3 and 4, participants will have the option to sign up to be a "vaccine ambassador," in which case they will get notifications when the study team posts new vaccine-related content, and will receive reminders about encouraging their friends to be vaccinated. The vaccine ambassadors will also be entered into a lottery to win prizes. The study team is building a website to host the videos of health professionals which answer common questions about Covid-19 vaccination. The investigators will measure engagement with the vaccine-related content as well as assess effects on vaccination rates at the county level.

DETAILED DESCRIPTION:
The study will have three treatment arms and a control group. Each of the treatments will be randomized at the county level and will be initiated through a Facebook ad campaign.

Experimental Sample: The experimental sample includes all states where less than 60% of the total population had received a first dose of Covid-19 vaccine by October 21, 2021. There are 1402 counties in the 19 states satisfying those criteria (Alabama, Alaska, Arkansas, Georgia, Idaho, Iowa, Indiana, Louisiana, Michigan, Mississippi, Missouri, Montana, North Dakota, Ohio, Oklahoma, South Carolina, Tennessee, West Virginia, Wyoming). Excluding the five counties with missing data, there are 1,397 counties in the experiment, of which there are 468 counties in the control group, 310 counties in T1 ("direct" messaging) treatment, 309 counties in T2 ("friends" messaging), and 310 counties in T3 ("gossips" messaging).

The following procedures will be used:

* Treatment Group 1 ("Direct" messaging): The investigators will conduct a Facebook ad campaign to show content about COVID-19 vaccination to a large number of Facebook users. Facebook will allocate ad credits across users in treatment areas. The ads will be displayed twice per week for 3-4 weeks. Like for any Facebook ad, individuals can choose to whether or not to watch the video and can close the ad at any time. If individuals wish, they can also share any of the content with others. The videos shown in the ads will be hosted on our project Facebook page "Doctors for Coronavirus Prevention." As in previous projects by the investigators, a health professional (normally wearing a white coat or scrubs) will read very short scripts directly onto the camera (see eg. https://www.facebook.com/doctors4covidprevention/posts/104965558099200 for an example).
* Treatment Group 2 ("Friends" messaging): For this group, the Facebook ad campaign will recruit individuals to become "vaccine ambassadors" to help spread the word about vaccination to their friends, families and communities. Recruitment ads will be disseminated in a similar manner to the content in T1. Individuals will be able to share the ad with others. Individuals interested in learning more can click through a link in the ad to the vaccine ambassador webpage. Participants can consume or share any of the information on the webpage. Interested individuals can also enroll formally as vaccine ambassadors. They can share their contact information with the study to a) be entered into prize lotteries, b) receive reminders to share content with others, c) be contacted in the future for possible follow-up surveys. They will be asked to give their informed consent at this time and will be screened based on whether they live in a treated county and whether they are 18 years or older.
* Treatment Group 3 ("Gossips" messaging): This treatment looks the same as Treatment Group 2, except the recruitment ads will differ slightly. If the individual clicks through to learn more about vaccine ambassadors, they will also be reminded to share the invitation with people they know who are often the source of important news or information.
* Control: individuals in these counties will receive no intervention and will never be contacted by members of the study team.

Treatment and control status at the county level will be merged with aggregated and de-identified datasets to measure COVID vaccinations, COVID symptoms, and cases, and engagement with the vaccine ambassador content.

The study team will create a series of websites with materials that the vaccine ambassadors can share with friends, family and others in their communities. This same content will be disseminated through sponsored Facebook ads in T1. On the website, the framing of the vaccine-related videos with either a "fact" or "myth" frame will be randomized. The purpose is to study which framing is more effective at engaging users.

ELIGIBILITY:
Inclusion Criteria:

* Facebook user
* Over 18 years old
* In a geographic area targeted by the study

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Duflo, PhD, Principal Investigator — Massachusetts Institute of Technology; Ben Olken, PhD, Principal Investigator — Massachusetts Institute of Technology; Abhijit Banerjee, PhD, Principal Investigator — Massachusetts Institute of Technology; Marcella Alsan, MD, PhD, Principal Investigator — Harvard Kennedy School; Arun Chandrasekhar, PhD, Principal Investigator — Stanford University; Emily Breza, PhD, Principal Investigator — Harvard University; Paul Goldsmith-Pinkham, PhD, Principal Investigator — Yale University; Emily Hoppe, PhD Student, Principal Investigator — Johns Hopkins School of Nursing; Pierre-Luc Vautrey, PhD Student, Principal Investigator — Massachusetts Institute of Technology; Lisa Ho, PhD Student, Principal Investigator — Massachusetts Institute of Technology; Lucy Ogbu-Nwobodo, MD, Principal Investigator — MGH/McLean Harvard Psychiatry Program; Erica Warner, ScD, MPH, Principal Investigator — Harvard Medical School & Massachusetts General Hospital; Carlos Torres, MD, Principal Investigator — Massachusetts General Hospital; Fatima Stanford, MD, MPH, MPA, Principal Investigator — Harvard Medical School & Massachusetts General Hospital; Sarah Eichmeyer, PhD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Massachusetts Institute of Technology, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share any individual participant data. The only individual participant data that the study will collect will be contact information through the "vaccine ambassador" program. "Vaccine ambassadors" are adults living in geographic areas assigned to Treatment 2 or Treatment 3 who have signed up on the study website to receive updates and reminders about vaccination-related content. However, the study team does not plan on collecting any information about the behavior of vaccine ambassadors, and so do not plan to share any of their data (which will just consisting of contact information) with other researchers.

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Counties
Groups:
- Treatment 2: Friends: Facebook users in the area receive ads which include videos of health professionals encouraging them to help their friends to get vaccinated. There is also a link in the ad to a website build by the study team. This website hosts videos which answer common questions about vaccination (the same videos which are directly served to Facebook users in Treatment 1).
  Doctor Videos: Receive ads on Facebook or through our website with videos in which health professionals tell people to get the Covid-19 vaccine. The health professionals answer common questions about the Covid-19 vaccine, such as how mRNA vaccines work, and what types of side effects to expect.
  Sharing Videos: Receive ads on Facebook with videos in which health professionals tell people to encourage their unvaccinated friends to get the Covid-19 vaccine.
  Vaccine Ambassador: Adults in participating geographic areas can sign up to be a "vaccine ambassador" on a website that the study team has built.
  Video framing: Visitors to the vaccine content website will randomly receive one framing of each video ("myth" or "fact").
  Video order: The order in which videos appear is randomized.
- Treatment 3: Gossips: Facebook users in the area receive ads which include videos of health professionals encouraging them to nominate their most influential friends to help their friends get vaccinated. The difference from Treatment 2 is that the health professionals call on Facebook users to get their most influential friends to do the convincing about the vaccine. There is also a link in the ad to a website built by the study team. This website hosts videos which answer common questions about vaccination (the same videos that are directly served to Facebook users in Treatment 1).
  Doctor Videos: Receive ads on Facebook or through our website with videos in which health professionals tell people to get the Covid-19 vaccine. The health professionals answer common questions about the Covid-19 vaccine, such as how mRNA vaccines work, and what types of side effects to expect.
  Sharing Videos (Influencers): Receive ads on Facebook with videos in which health professionals tell people to get their most influential friends to encourage their unvaccinated friends to get the Covid-19 vaccine.
  Vaccine Ambassador: Adults in participating geographic areas can sign up to be a "vaccine ambassador" on a website that the study team has built.
  Video framing: Visitors to the vaccine content website will randomly receive one framing of each video ("myth" or "fact").
  Video order: The order in which videos appear is randomized.
Period: Overall Study
Arm/Group | Control | Treatment 1: Direct | Treatment 2: Friends | Treatment 3: Gossips
Started (The number of participants in each group is the number of people who signed up as a "vaccine ambassador" in each treatment arm. The Facebook ads were not run in control group counties.) | NA; 417 Counties (Vaccine Ambassadors were not enrolled in the control group.) | NA; 275 Counties (5933089 unique Facebook users saw the study's Treatment 1 (Direct) social media campaign. Vaccine Ambassadors were not enrolled in the Treatment 1: Direct arm.) | 4; 274 Counties (5952765 unique Facebook users saw the study's Treatment 2 (Friends) social media campaign.) | 2; 276 Counties (5942915 unique Facebook users saw the study's Treatment 3 (Gossips) social media campaign.)
Completed (The study intervention was a social media campaign that displayed ads on Facebook which encouraged people to get a Covid-19 vaccine. As there was no way to "complete" the study, the number of participants who started and the number of participants who completed the study is the same.) | NA; 417 Counties (417 counties were randomized to the control group, where no social media campaign was served. No intervention was carried out in the control group, and the only data used were publicly available county-level data. Vaccine Ambassadors were not enrolled in the Treatment 1: Direct arm.) | NA; 275 Counties (Vaccine Ambassadors were not enrolled in the Treatment 1: Direct arm.) | 4; 274 Counties | 2; 276 Counties
Not Completed | NA; 0 Counties | NA; 0 Counties | 0; 0 Counties | 0; 0 Counties

BASELINE CHARACTERISTICS:
Population: The analysis used publicly available county-level data, and so the baseline variables all had county-level granularity. We did not collect any person-level baseline measures.
Units Other Than Participants: Counties
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Treatment 1: Direct | Treatment 2: Friends | Treatment 3: Gossips | Total
Number analyzed (Participants) | NA | NA | NA | NA | NA
Number analyzed (Counties) | 417 | 275 | 274 | 276 | 1242
Age, Customized [Number; unit: participants] — Population: Age data not collected
  participants
    number analyzed (Counties) | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: percent] — Population: Gender data was not collected. All gender data used were publicly available county-level data that was not collected for this experiment. We do not collect individual-level baseline data.
  percent
    number analyzed (Counties) | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Units; unit: Counties] — Ethnicity data not collected Population: Ethnicity data not collected
  Counties
    number analyzed (Counties) | 0 | 0 | 0 | 0 | 0
    Hispanic or Latino |  |  |  |  | 0
    Not Hispanic or Latino |  |  |  |  | 0
    Unknown or Not Reported |  |  |  |  | 0
Race (NIH/OMB) [Count of Units; unit: Counties] — Population: Race data not collected
  Counties
    number analyzed (Counties) | 0 | 0 | 0 | 0 | 0
    American Indian or Alaska Native |  |  |  |  | 0
    Asian |  |  |  |  | 0
    Native Hawaiian or Other Pacific Islander |  |  |  |  | 0
    Black or African American |  |  |  |  | 0
    White |  |  |  |  | 0
    More than one race |  |  |  |  | 0
    Unknown or Not Reported |  |  |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in County-Level Covid-19 Vaccination Measured by Inverse Hyperbolic Sine
Description: County-level Covid-19 vaccination rates were analysed using publicly available data. The number of new vaccinations in each county was transformed using the inverse hyperbolic sine because the underlying vaccination count data were right-skewed and included zeros. Larger numbers are considered better in the context of the study (more people vaccinated).
Time Frame: During intervention (6 weeks) and after intervention (3 weeks)
Population: Counties were randomized into treatment groups, and outcome data are public county-level data.
Measure: Mean (95% Confidence Interval); unit: asinh(new dose 1s of vaccine)
Units Other Than Participants: Counties
Arm/Group | Control | Treatment 1: Direct | Treatment 2: Friends | Treatment 3: Gossips
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (Counties) | 417 | 275 | 274 | 276
asinh(new dose 1s of vaccine) | 0 [0 to 0] | -0.023 [-0.10 to 0.055] | -0.007 [-0.081 to 0.067] | -0.037 [-0.11 to 0.034]

ADVERSE EVENTS:
Description: As the treatment was a social media campaign administered on Facebook, and individual-level information was not collected for people who simply watched the ads, the study could not monitor for adverse events. "Vaccine ambassadors" were also not monitored for adverse events, as their risk from the study was very small (the only additional interaction between the study and "vaccine ambassadors" was to contact one participant who had won a gift card.)
Arm/Group | Control | Treatment 1: Direct | Treatment 2: Friends | Treatment 3: Gossips
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT05182554/Prot_SAP_000.pdf